CLINICAL TRIAL: NCT04352920
Title: Vacuum Myofascial Therapy Device in Treatment of Muscle Fibrosis
Acronym: Physium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Manuel Rodriguez Huguet, Clinical Professor, University of Cadiz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27/19
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Muscle Injury
Keywords: negative pressure; cupping; physical therapy modalities

STUDY DESIGN:
Intervention Model Description: Medical Doctor diagnosed muscle fibrosis
Masking Description: Outcomes assesor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): PHYSIUM System® provides standardized negative pressure massage for 15 minutes with the analgesic program and 15 minutes with the trigger points program at 80 millibars with eight adjustable arms both in the entire muscle and in muscle fibrosis.
  Interventions: Other: Experimental group

INTERVENTIONS:
Other: Experimental group — PHYSIUM System® provides standardized negative pressure massage for 15 minutes with the analgesic program and 15 minutes with the trigger points program at 80 millibars with eight adjustable arms both in the entire muscle and in muscle fibrosis.

SUMMARY:
We present the case of a 24-year-old professional soccer player, with no personal history of interest, who came to the X-Ray diagnosis service due to severe pain in the right quadriceps muscle after a 10-month evolution of muscle rupture occurred during sports practice.

DETAILED DESCRIPTION:
PHYSIUM System® provides standardized negative pressure massage for 15 minutes with the analgesic program and 15 minutes with the trigger points program at 80 millibars with eight adjustable arms, both in the entire muscle and in muscle fibrosis.

Seven days later, after PHYSIUM System® session with the same parameters of the previous treatment, ultrasound elastography was performed.

ELIGIBILITY:
Inclusion criteria.

* 24-year-old professional soccer player.
* No personal medical history of interest

Min Age: 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
The intensity of pain in muscle fibrosis | Baseline
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of elbow pain, and the worst and lowest level of pain experienced in the preceding week.

SECONDARY OUTCOMES:
The intensity of pain in muscle fibrosis | Two weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of elbow pain, and the worst and lowest level of pain experienced in the preceding week.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Rodriguez Huguet, Physiotherapy, Principal Investigator — University of Cádiz
Locations (1):
- Manuel Rodríguez Huguet, Cadiz, Cádiz, Spain

REFERENCES:
- [Result] Bhatia K, Tong CS, Cho CC, Yuen EH, Lee J, Ahuja AT. Reliability of shear wave ultrasound elastography for neck lesions identified in routine clinical practice. Ultraschall Med. 2012 Oct;33(5):463-8. doi: 10.1055/s-0032-1325330. Epub 2012 Oct 15. PMID 23070932
- [Result] Ekstrand J, Askling C, Magnusson H, Mithoefer K. Return to play after thigh muscle injury in elite football players: implementation and validation of the Munich muscle injury classification. Br J Sports Med. 2013 Aug;47(12):769-74. doi: 10.1136/bjsports-2012-092092. Epub 2013 May 5. PMID 23645834
- [Result] Hallen A, Ekstrand J. Return to play following muscle injuries in professional footballers. J Sports Sci. 2014;32(13):1229-36. doi: 10.1080/02640414.2014.905695. Epub 2014 May 1. PMID 24784885
- [Result] Fousekis K, Tsepis E, Poulmedis P, Athanasopoulos S, Vagenas G. Intrinsic risk factors of non-contact quadriceps and hamstring strains in soccer: a prospective study of 100 professional players. Br J Sports Med. 2011 Jul;45(9):709-14. doi: 10.1136/bjsm.2010.077560. Epub 2010 Nov 30. PMID 21119022